CLINICAL TRIAL: NCT07126275
Title: Mirror Journaling App Study
Acronym: Mirror Journal
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Mind Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080718
Record Dates: First submitted 2025-02-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Depression Symptoms; Anxiety Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mirror Guided Journaling + Mood Tracking (Experimental): Structured prompts and regular feedback to facilitate journaling, alongside daily mood tracking in the Mirror App.
  Interventions: Device: Mirror App Journaling and Mood Tracking Study
- Mirror Unguided Journaling + Mood Tracking (Experimental): Free-form journaling with access to daily mood tracking in the Mirror app without specific guided prompts.
  Interventions: Device: Mirror App Journaling and Mood Tracking Study
- Mirror Mood Tracking Only (Experimental): Daily mood tracking in the Mirror app, without any journaling component.
  Interventions: Device: Mirror App Journaling and Mood Tracking Study
- Control Group (No Intervention): Information on mental health resources without journaling or mood tracking.

INTERVENTIONS:
Device: Mirror App Journaling and Mood Tracking Study — Mirror is a mobile journaling app developed by the Child Mind Institute (CMI) for youth who want to explore and improve their mental health, particularly addressing symptoms related to depression. The Mirror app enables users to express their thoughts and emotions through multimodal entries (i.e., written, voice, selfie video) and provides prompts to facilitate journal entries using unique, emotionally supportive features to help users identify and process emotions. Users can also complete free-form, unguided journaling, and can complete daily mood tracking and see changes/progress over time.
  Arms: Mirror Guided Journaling + Mood Tracking; Mirror Mood Tracking Only; Mirror Unguided Journaling + Mood Tracking

SUMMARY:
This study has three primary aims: 1) Validate Mirror's Mood Check feature by measuring convergent validity;2) Assess user experience and acceptability metrics (e.g., usability, engagement, satisfaction) of the Mirror app, with a particular focus on the journaling feature; 3) Assess the impact of guided journaling and mood tracking on depressive and anxious symptoms.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Depression is a common and serious mental disorder that can negatively affect an individual's thoughts, feelings, and ability to perform daily activities. The onset of depression can occur at any stage of life. The estimated prevalence of depression in childhood is low (1.09%) and the highest in young adulthood (21%) , with a sharp increase seen during adolescence . In 2022, 15.08% of adolescents between the ages of 12 and 17 reported suffering from at least one major depressive episode in the past year. Of those, only 27.2% received consistent treatment. Depression in adolescents, particularly if left untreated, is associated with negative consequences later in life, such as higher levels of substance use disorders, worse health and social functioning, less educational and financial achievement, and increased criminality. Considering these serious and lasting consequences, depression in adolescents is a significant public health issue that deserves proactive approaches to prevent or mitigate its negative impact on individuals and society.

Journaling is recognized as a common, non-pharmacological tool in the management of mental disorders, including depression. Journaling can promote self-reflection and self-awareness, which can help improve mental health (e.g., enhance emotional regulation, reduce stress, facilitate behavioral changes). Although digital journaling can offer equivalent expression and release as traditional journaling with pen and paper, digital journaling has many advantages, such as enhanced accessibility, data organization, data security, analytic potential, and multimedia integration; these features make digital journaling a highly efficient tool for managing mental health. As such, a growing body of research supports the clinical benefits of digital journaling for depression in adults. Yet, the acceptability and efficacy of digital journaling in adolescents are understudied, calling for further investigation.

Mirror is a mobile journaling app developed by the Child Mind Institute (CMI) for youth who want to explore and improve their mental health, particularly addressing symptoms related to depression. Like other mobile journaling apps, the Mirror app enables users to express their thoughts and emotions through multimodal entries (i.e., written, voice, selfie video) and provides prompts to facilitate journal entries. However, the Mirror app offers unique, emotionally supportive features to help users identify and process emotions. First, Mirror users can explore multimodal guided journaling (e.g., video, audio, and written entries with guided prompts); as the app's name suggests, one of the guides encourages users to stand in front of a mirror and start video journaling while making eye contact with themselves. This guided journaling using a mirror can help increase users' self-reflection and self-expression. Second, the Mirror app has a user-centered mood-checking feature ("Mood Check") designed based on the circumplex model of emotions, in which the x- and y-axis represent pleasantness and energy level, respectively. Mirror's Mood Check feature is visually appealing (i.e., two sliders corresponding to the two axes) and allows users to gain more granular insights into their emotional states.

With these unique and user-centered features described above, the Mirror app has great potential for increasing adolescent users' engagement, which could significantly influence the efficacy of digital journaling on mental health. Importantly, the information gained from the proposed study will guide the development of future clinical trials for adolescents suffering from depression.

PROPOSED STUDY

This study has three primary aims: 1) Validate Mirror's Mood Check feature by measuring convergent validity;2) Assess user experience and acceptability metrics (e.g., usability, engagement, satisfaction) of the Mirror app, with a particular focus on the journaling feature; 3) Assess the impact of guided journaling and mood tracking on depressive and anxious symptoms.

This study will enroll 500 young adults ages 18-25 via Prolific Academic (https://www.prolific.com/) an online research participant recruitment tool.

Users on Prolific Academic must be the age of majority in the locality in which they register for an account. Prolific users ages 18-25 that reside in the U.S., have access to a smart device, and are willing to download an external app (screened by Prolific Academic), will be eligible to complete a screening form. Participants with mild to moderate depressive or anxiety symptoms will be eligible to enroll in the study.

Participants on Prolific will complete a baseline assessment and will then be randomized to complete one of four study conditions over the course of 8 weeks:

1. Guided Journaling + Mood Tracking: Structured prompts and regular feedback to facilitate journaling, alongside daily mood tracking.
2. Unguided Journaling + Mood Tracking: Free-form journaling with access to mood tracking tools without additional guidance.
3. Mood Tracking Only: Mood tracking tools without any journaling component.
4. Control Group: Information on mental health resources without journaling or mood tracking.

In addition to their journaling and mood check assignments, all participants will also complete a weekly check in questionnaire, post-study and one month follow up assessment of symptoms and user satisfaction with the app.

ELIGIBILITY:
Inclusion Criteria:

* Prolific users ages 18-25
* Must reside in the U.S.
* Must have access to a smart device, and are willing to download an external app (screened by Prolific Academic)
* Must complete screening form which consists of the Patient Health Questionnaire (PHQ-2) and the Generalized Anxiety Disorder (GAD-7) Scale.
* Must have mild to moderate depressive or anxiety symptoms, as measured by the screening form

Exclusion Criteria:

- None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | 12 weeks (including 1 month follow up)
  Statistical models including ANOVA and regression will be used to compare changes in depressive symptoms across the four groups. Changes in depressive symptoms will be assessed with the Patient Health Questionnaire 8 item (PHQ-8), which has scores that range from 0-24 with higher scores indicating higher levels of depressive symptoms.
  Depressive Symptoms will be measured at baseline, post 8-weeks of the intervention, and at a 1 month follow up.
Anxiety Symptoms | 12 weeks (including 1 month follow up)
  Statistical models including ANOVA and regression will be used to compare changes in anxiety symptoms across the four groups. Changes in anxiety symptoms will be assessed with the Generalized Anxiety Disorders Scale (GAD-7), which has scores that range from 0-24 with higher scores indicating higher levels of anxiety symptoms.
  Anxiety Symptoms will be measured at baseline, post 8-weeks of the intervention, and at a 1 month follow up.
Impairment | 12 weeks (including 1 month follow up)
  Statistical models including ANOVA and regression will be used to compare changes in impairment across the four groups. Changes in impairment will be assessed with the WHO Disability Assessment Schedule (WHODAS 2.0), which has scores that range from 0-100 with higher scores indicating higher levels of impairment.
  Impairment will be measured at baseline, post 8-weeks of the intervention, and at a 1 month follow up.

SECONDARY OUTCOMES:
User Experience | 8 weeks
  User experience data will also be collected and analyzed to support product improvement. Data will be collected with the The MAUQ, or mHealth App Usability Questionnaire, a tool used to assess the usability of mobile health (mHealth) applications. It provides a structured way to gather user feedback and determine how easy and useful an app is for its intended purpose using likert scale questions.
User Experience | 8 weeks
  User experience data will be collected and analyzed to support product improvement. Data will be collected with the System Usability Scale (SUS), a ten-item Likert scale giving a global view of subjective assessments of usability, which generates a score from 0-100 with higher scores indicating higher levels of usability.
User Feedback | 8 weeks
  User experience data will be collected and analyzed to support product improvement. Data will be collected with a feedback questionnaire developed by the Child Mind Institute that asks questions specifically about the Mirror platform. The assessment includes both close and open ended questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milham, MD, PhD, Principal Investigator — Child Mind Institute
Locations (1):
- Child Mind Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No